CLINICAL TRIAL: NCT00001190
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial of Luteinizing Hormone-Releasing Hormone Analog (LHRHa) in Pubertal Patients With Extreme Short Stature
Brief Title: Study of Luteinizing Hormone-Releasing Hormone Analog (LHRHa) in Pubertal Patients With Extreme Short Stature
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 830199; 83-CH-0199
Record Dates: First submitted 1999-11-03; First posted 2002-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-10

CONDITIONS: Dwarfism; Growth Disorder
Keywords: Growth; Adolescence; Children
MeSH Terms: conditions — Dwarfism; Growth Disorders | interventions — deslorelin

INTERVENTIONS:
Drug: Deslorelin

SUMMARY:
Children with extreme short stature (height) and their families often experience significant psychological stress related to concerns about adult height. In addition, short stature often results in life-long emotional, social, and physical obstacles to the affected person.

Normal growth occurs in two phases. The first phase, known as childhood growth, occurs below the age of 10. The second phase of growth, teen-age or adolescent growth, begins between the ages of 10 and 15. In addition, puberty marks the time when the bone's growth plates (epiphysis) begin to close, initiating the completion of linear growth (height).

Some children suffer from a condition called precocious puberty, meaning that puberty begins at a younger age than normal. The development of medications known as synthetic LHRH analogs have provided a method to delay puberty and treat these patients.

LHRHa (deslorelin) is a hormone created to act like naturally occurring LHRH. It been used in patient's diagnosed with precocious (early onset) puberty. The drugs were able to regress patient's clinical signs of puberty, decrease the levels of adult sex hormones produced, and slow the rate of bone aging.

DETAILED DESCRIPTION:
Children with extreme short stature and their families frequently experience significant psychological stress related to concerns about adult height. Additionally, extreme short stature often presents life-long emotional, social, and physical obstacles to the affected individual. The onset of puberty in such patients presents a critical management problem because puberty initiates the process of epiphyseal closure that terminates linear growth. Until recently, there was no way to delay the onset of puberty in such patients. The development of synthetic LHRH analogs, however, has provided such a method. Administration of such analogs to children with precocious puberty caused a regression of their clinical signs of puberty, a decrease in their gonadotropins and sex steroids, and a slowing of the rate of bone age advancement.

We propose to treat pubertal children with extreme short stature with a long-acting analog of luteinizing hormone-releasing hormone (D-Trp6-Pro9-NEt-LHRHa). The goal of LHRHa treatment in these children is to halt the normal progression into puberty and thereby delay epiphyseal fusion. We postulate that delay of puberty will prolong pre-pubertal growth prior to the pubertal spurt and subsequent epiphyseal fusion, and thus will enhance ultimate height. This study will test this hypothesis through a double-blind, randomized comparison of the effect of LHRHa and placebo on final adult height. Patients will be treated with LHRHa or placebo for 4 years, and will then be followed until they have completed puberty and have stopped growing.

ELIGIBILITY:
Patients with extreme short stature will qualify for inclusion under this protocol if they meet the following criteria:

Age 9 through 15.99 years at the start of treatment.

Tanner II-V pubertal development.

Height at least 2.25 S.D. below the median for chronologic age at the time of pubertal onset, or a predicted adult height at least 2.25 S.D. below median adult height.

The height criterion must be met before study entry, but not necessarily on the actual date the patient starts to take the protocol injections because advancing puberty may cause an increase in height velocity that temporarily increases height standard deviation score.

Unfused carpal and phalangeal epiphyses by bone age x-ray.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1983-11; Study Completion 2001-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Municchi G, Rose SR, Pescovitz OH, Barnes KM, Cassorla FG, Cutler GB Jr. Effect of deslorelin-induced pubertal delay on the growth of adolescents with short stature and normally timed puberty: preliminary results. J Clin Endocrinol Metab. 1993 Nov;77(5):1334-9. doi: 10.1210/jcem.77.5.8077329.
- [Background] Manasco PK, Pescovitz OH, Hill SC, Jones JM, Barnes KM, Hench KD, Loriaux DL, Cutler GB Jr. Six-year results of luteinizing hormone releasing hormone (LHRH) agonist treatment in children with LHRH-dependent precocious puberty. J Pediatr. 1989 Jul;115(1):105-8. doi: 10.1016/s0022-3476(89)80341-5. No abstract available. PMID 2661787
- [Background] Bourguignon JP. Linear growth as a function of age at onset of puberty and sex steroid dosage: therapeutic implications. Endocr Rev. 1988 Nov;9(4):467-88. doi: 10.1210/edrv-9-4-467. No abstract available. PMID 3065075